CLINICAL TRIAL: NCT04783246
Title: Feasibility and Effectiveness of a Virtual Group Fitness and Nutrition Intervention in Individuals With Psychosis: A Pilot Study
Brief Title: Virtual Group Fitness and Nutrition Intervention for Individuals With Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H-40042
Record Dates: First submitted 2021-02-28; First posted 2021-03-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia Spectrum Disorder (SSD)
Keywords: Lifestyle changes; Fitness instruction; Nutrition education; Virtual interventions
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A two-period cross over design will be implemented to compare between groups in a self-paired manner to minimize the effects of confounding covariates. Participants will agree to either immediate randomization to the non-intervention period or the intervention period at the time of consent. Participants will be randomized utilizing conceal block randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- Intervention/Non-Intervention (Experimental): Participants in this arm will initially be randomized to the intervention period and will receive the interventions for 11 weeks followed by no interventions for 11 weeks.
  Interventions: Behavioral: Group Fitness; Other: Nutrition education
- Group B- Non-Intervention/Intervention (Active Comparator): Participants in this arm will initially be randomized to the non-intervention period for 11 weeks followed by the intervention period for 11 weeks.
  Interventions: Behavioral: Group Fitness; Other: Nutrition education

INTERVENTIONS:
Behavioral: Group Fitness — The group fitness intervention will involve streaming a group fitness class lead by a certified personal trainer. certified personal trainer and include variations of body-weight strength and aerobic exercise activities. Each work out session will be 30 minutes in duration and follow a structure of a warm-up period, alternating strength and aerobic exercises of varying intensity, and a cool-down period. The videos will be streamed to the group by a facilitator over Zoom video conferencing.
Other: Nutrition education — The nutrition education intervention will involve 45-minute educational sessions involving didactic teaching, interactive goal setting, and a live cooking demonstration. Each session will be taught by a registered dietician who will also be responsible for designing the curriculum schedule.

SUMMARY:
Individuals with schizophrenia spectrum disorder (SSD) often face unique barriers that limit the development of long-lasting lifestyle changes. In this study, The investigators will investigate the feasibility and impact of a novel lifestyle intervention in individuals with schizophrenia or schizoaffective disorder. The intervention will be composed of group fitness instruction and educational nutrition didactics that will be accessible to participants at-home through remote streaming. The fitness component will consist of weekly group fitness sessions delivered by a certified personal trainer over a virtual interface. The educational nutritional component of this intervention will involve interactive didactic sessions designed to improve knowledge of nutrition and positively change dietary behavior in this population.

ELIGIBILITY:
Inclusion Criteria:

* Receiving outpatient psychiatric care for early-episode psychosis, schizophrenia, or schizoaffective disorder at Boston Medical Center or the Mass General Hospital
* Proficient in English
* Cleared by their primary care provider to perform 30 minutes of aerobic and strength exercise

Exclusion Criteria:

* Documented history of one of the absolute contraindications to exercise defined in the "Exercise Standards for Testing and Training" by the American Heart Association in our electronic medical record which includes the following:

  1. Acute myocardial infarction
  2. Ongoing unstable angina
  3. Uncontrolled cardiac arrhythmia with hemodynamic compromise
  4. Endocarditis
  5. Symptomatic severe aortic stenosis
  6. Decompensated heart failure
  7. Acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis
  8. Acute myocarditis or pericarditis
  9. Acute aortic dissection
* Inability to ambulate independently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Feasibility of lifestyle intervention | 22 weeks
  Feasibility of the lifestyle intervention will be assessed by the satisfaction level of participants which will be obtained from questions on an investigator developed questionnaire. Higher satisfaction levels will suggest greater feasibility.
Tolerability of educational nutritional sessions | 22 weeks
  Individual attendance levels will be measured at weekly intervals during educational nutrition didactic sessions. Attendance will be calculated as the total number of attended groups divided by the total number of eligible groups to account for the late enrollment of individuals.
Tolerability of group fitness classes | 22 weeks
  Individual attendance levels will be measured at weekly intervals during group fitness classes. Attendance will be calculated as the total number of attended groups divided by the total number of eligible groups to account for the late enrollment of individuals.

SECONDARY OUTCOMES:
Change in physical activity level | baseline, 22 weeks
  Change in physical activity level will be measured through step counts which will be collected throughout the active intervention period via pedometers provided to study participants at the beginning of the trial period. Step counts will be logged weekly at group fitness classes.
Change in weight | baseline, 22 weeks
  Participants will be asked to weigh themselves and document their weight. Either before or after each session the participant will share their weight with a research assistant on a phone call without other participants present.
Change in resting heart rate | baseline, 22 weeks
  Participants will be taught how to obtain a resting heart rate and asked to document their resting heart rate. Either before or after each session the participant will share their resting heart rate with a research assistant on a phone call without other participants present.
Change in Hemoglobin A1c level (HbA1c) | baseline, 22 weeks
  Study staff will abstract the HbA1c levels from the patient's Boston Medical Center (BMC) electronic record.
Change in psychological well being | baseline, 22 weeks
  Change in psychological well-being will be assessed through the administration of the Personal Health Questionnaire-9 (PHQ-9).The PHQ-9 has been previously validated in the general population to assess for major depressive disorder and subclinical depressive symptoms. Scores can range from 1-27 and the higher the score the greater the depressive symptoms.
Change in self esteem | baseline, 22 weeks
  The change in scores from baseline to 22 weeks from the 12-item Short Form Health Survey (12-SFHS), State Self-Esteem Scale (SSES) will be used to assess self esteem change. The SSES scale has been validated in multiple populations as an assessment of an individual's sense of worthiness in three domains: (1) appearance, (2) performance, and (3) social Each item is scored on a 5-point scale (1 = not at all, 2 = a little bit, 3 = somewhat, 4 = very much, and 5 = extremely). Scores range form 20 to 100 and higher scores are associated with higher self esteem.
Change in psychotic episodes | baseline, 22 weeks
  Change in psychotic symptoms will be assessed through implementation of the Brief Psychiatric Rating Scale (BPRS). The BPRS is a validated instrument which measures several constructs important to the assessment of the severity of symptoms of psychosis such as degree of hallucinations, unusual thought content, self-neglect, and conceptual disorganization. Higher scores are associated with more psychotic episodes
Motivation to exercise | 22 weeks
  Change in motivation to exercise will be measured through administration of Behavioral Regulation Exercise Questionnaire-3 (BREQ-3). Higher scores are associated with greater motivation to exercise.
Change in nutritional knowledge | baseline, 22 weeks
  Change in nutrition knowledge will be measured through comparison of baseline and post intervention multiple choice test written by a registered dietician.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Brown, MD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No